CLINICAL TRIAL: NCT00359476
Title: A Multicenter, Single-Arm, Phase II Study of Single-Agent Vinflunine in the Second-line Treatment of Patients With Gastric Cancer
Brief Title: A Study of Vinflunine in Patients With Gastric Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA183-023
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-12

CONDITIONS: Stomach Cancer
Keywords: Locally advanced/metastatic gastric adenocarcinoma; adenocarcinoma-gastroesophageal junction; Gastric Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Vinflunine

INTERVENTIONS:
Drug: Vinflunine — solution for injection, IV, 280/320 mg/m2, every 3 wks, variable duration

SUMMARY:
The purpose of this study is to learn if vinflunine can shrink or slow the growth of cancer in patients with advanced or metastatic stomach cancer who have progressed on a prior treatment with a fluoropyrimidine or taxane-containing chemotherapy regimen. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic gastric adenocarcinoma, including adenocarcinoma of the gastroesophageal junction who have progressed on a fluoropyrimidine or taxane-containing regimen in any combination in one prior first line treatment.
* EGOC performance status of 0,1 or 2
* Men and women, 18 years of age and older

Exclusion Criteria:

* Patients having received more than one previous systemic chemotherapy regimen in any setting.
* Major abdominal surgery within 2 months or any other surgery under general anesthesia within 4 weeks
* Unresolved occlusive or sub-occlusive intestinal disease or any significant chronic intestinal disease (e.g. ulcerative colitis)
* Prior radiation to >=30% of the bone marrow and/or radiation within 4 weeks prior to enrollment
* Acute or chronic hepatitis
* Known HIV infection
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms
* A history of additional risk factors for Torsade de Pointes (e.g., heart failure hypokalemia, family history of Long QT Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The Response Rate (RR: Complete Response [CR]+Partial Response [PR], as defined by Response Evaluation Criteria in Solid Tumors [RECIST] | throughout the study

SECONDARY OUTCOMES:
Estimation of the progression free survival and overall survival | At the end of the study
The estimation of the disease control rate | At the end of the study
The time to response and the duration of response | At the end of the study
The evaluation of the safety profile of vinflunine | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Local Institution, Kampung Baharu Nilai, Negeri Sembilan, Malaysia
- Local Institution, Quezon City, Philippines
- South Korea (3):
  - Local Institution, Suwon, Gyeonggi-do
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul